CLINICAL TRIAL: NCT04278742
Title: A Collaborative Approach in Diabetes Foot Education - A Pragmatic Randomised Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGH_collab_edu
Record Dates: First submitted 2018-12-17; First posted 2020-02-20 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2; Neuropathy;Peripheral
Keywords: patient education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Neuritis | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Suitable participants recruited and randomised into Study Intervention Group or Control Group.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional - collaborative education (Experimental): Collaborative style of communication whereby the clinician and patient co-creates the treatment plan
  Interventions: Other: Patient education
- Control group (No Intervention): Traditional directive and didactic style of patient information will be provided

INTERVENTIONS:
Other: Patient education — Using a collaborative approach to engage patients in their own care, allowing patients to continue to have full control of their treatment. The clinician and patient co-creates the treatment plan.
  Other Names: Collaborative counselling
  Arms: Interventional - collaborative education

SUMMARY:
Traditional directive style of requesting or demanding compliance to set behavior is found to have little effect on patient's self-care behavior. It is reported that patients prefer to restate or rephrase their understanding in a care setting, instead of a directive/didactic approach where the clinician provides 'one-way' information. In fact, directive persuasion is thought to lead to resistance to change and is counter-effective.

New approaches such as open ended communication, interview style and collaborative approach is found to engage patients better in their own care and elicit patient's own intrinsic motivations for making changes. One way to do this is to

1. invite patient to share their thoughts or concerns then
2. clarify patient's understanding

From their responses:

(3a) affirm patient's correct understanding or (3b) address misconceptions with permission.

In this study, the investigators will randomize 240 subjects into two groups: Group A will undergo the above describe collaborative approach to patient education and counselling; Group B will undergo current (traditional, didactic approach) patient education. It is hypothesized that the collaborative approach group (Group A) should experience better understand of their health condition and foot ulcer, be better able to adhere to treatment plan through collaborative participation and overall be more satisfied with the treatment. Outcomes will be tracked at (i) post intervention and (ii) 4 months post intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed type II diabetes
2. Above age 21
3. Plantar foot ulcer - high risk with active full-thickness ulcer
4. Pedal pulses palpable or min toe pressure of 30mmHg
5. Medium of language: English
6. Activities of daily living (ADL) independent (without carer)

Exclusion Criteria:

1. Diagnosed mental health conditions
2. Diagnosed cognitive impairment
3. Diagnosed visual impairment
4. Diagnosed hearing and speech disabilities

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Wound healing | 12 weeks
  Percentage patients with healed wound (wound size = 0cm)

SECONDARY OUTCOMES:
Knowledge score assessed by questionnaire | Week 1 and week 12
  Knowledge score in Knowledge & Behaviour questionnaire (Maximum score 16)
Behaviour score assessed by questionnaire | Week 1 and week 12
  Behaviour score in Knowledge & Behaviour questionnaire (Maximum score 59)

CONTACTS AND LOCATIONS:
Overall Officials: Marabelle Heng, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be available to the PI. The study team will be analysing de-identified data

REFERENCES:
- [Background] Gabbay RA, Kaul S, Ulbrecht J, Scheffler NM, Armstrong DG. Motivational interviewing by podiatric physicians: a method for improving patient self-care of the diabetic foot. J Am Podiatr Med Assoc. 2011 Jan-Feb;101(1):78-84. doi: 10.7547/1010078. PMID 21242475
- [Background] Kemp EC, Floyd MR, McCord-Duncan E, Lang F. Patients prefer the method of "tell back-collaborative inquiry" to assess understanding of medical information. J Am Board Fam Med. 2008 Jan-Feb;21(1):24-30. doi: 10.3122/jabfm.2008.01.070093. PMID 18178699